CLINICAL TRIAL: NCT04503876
Title: Pulmonary and Ventilatory Effects of End-expiratory Positive Pressure Optimization in Intubated ICU Patients With Healthy Lungs or Acute Respiratory Distress Syndrome. A Randomized Controlled Trial
Brief Title: Effects of End-expiratory Positive Pressure Optimization in Intubated Patients With Healthy Lung or Acute Respiratory Distress Syndrome
Acronym: PEEP-Réa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RBHP 2019 GODET (Peep Réa)
Record Dates: First submitted 2020-07-13; First posted 2020-08-07 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: ICU Patients; Healthy Lung; Positive End-Expiratory Pressure; ARDS; Alveolar Recruitment Maneuver
Keywords: ICU patients; Volume-controlled ventilation; Open lung strategy; PEEP titration; Alveolar recruitment maneuver; ARDS; Healthy lungs; Intubation; Tracheotomy; End-expiratory lung volume; Electro-impedance tomography; Recruited lung volume

STUDY DESIGN:
Intervention Model Description: Interventional trial comparing two strategies of PEEP optimization during mechanical ventilation in two groups of ICU patients: with healthy lungs or with ARDS. The study consists of comparing pulmonary pathophysiological parameters for different PEEP levels. The first strategy implies the use of an ARM followed by a stepwise decremental PEEP titration whereas the second considers a stepwise incremental PEEP titration without any previous ARM, during controlled invasive mechanical ventilation. Each patient will receive both strategies in a random consecutive order
Who Masked: Participant
Masking Description: Statistical analysis will be conducted by an independant statistician not involved in data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Decremental PEEP titration following an ARM (Active Comparator): PEEP will be titrated in a stepwise decremental fashion following a standardized alveolar recruitment maneuver (ARM). The ARM is a progressive increase of intra-thoracic pressure (pressure controlled mode), with a constant driving pressure of 10 cmH2O and PEEP steps (10-15-20-25-30-35 and 40 cmH2O), reaching a maximum pressure of 50 cmH2O, allowing full recruitment. PEEP steps will be conducted every 2 cmH2O (from 20 to 6 cmH2O), every 5 minutes.
  Interventions: Other: Decreasing PEEP setting
- Incremental PEEP titration without any previous ARM (Active Comparator): PEEP will be titrated in a stepwise incremental fashion without any previous alveolar recruitment maneuver (ARM). PEEP steps will be conducted every 2 cmH2O (from 6 to 20 cmH2O), every 5 minutes.
  Interventions: Other: Increasing PEEP setting

INTERVENTIONS:
Other: Increasing PEEP setting — End expiratory lung volume and lung aeration measurements will be conducted using electrical impedance tomography and nitrogen washin-washout method. Measurements will be conducted during the last minute of each step.
  Arms: Incremental PEEP titration without any previous ARM
Other: Decreasing PEEP setting — End expiratory lung volume and lung aeration measurements will be conducted using electrical impedance tomography and nitrogen washin-washout method. Measurements will be conducted during the last minute of each step.
  Arms: Decremental PEEP titration following an ARM

SUMMARY:
PEEP titration is a recommended during invasive mechanical ventilation of ICU patients. However, little is known about the right way to conduct this titration. PEEP titration can be conducted by a stepwise increase in PEEP level, or following an ARM and a consecutive stepwise decrease in PEEP level. Those 2 methods will be explored in intubated ICU patients either with healthy lung or ARDS lungs. Physiological exploration will include end-expiratory lung volume measurements, driving pressure, compliance and electro-impedance tomography at each PEEP level.

DETAILED DESCRIPTION:
Management of ICU patients may require the use of ventilatory support requiring tracheal intubation and invasive mechanical ventilation.

Any mechanically ventilated patient is exposed to the formation of atelectasis (collapsed pulmonary alveoli), which occurs systematically after endotracheal tube insertion, after any de-recruiting action (tracheal suction, disconnection) or simply if protective ventilation is used, combining small tidal volumes (6 to 8 mL/kg of theoretical ideal body weight - IBW) and an end-expiratory positive pressure (PEEP) that is sometimes insufficient. It is thus proposed to perform alveolar recruitment maneuvers (ARMs), which remove atelectasis by temporarily increasing intrathoracic pressure. To avoid alveolar re-collapse, it is necessary to apply a sufficient level of PEEP.

The opening pressure (P) necessary for the re-expansion of a collapsed alveolus is inversely proportional to its radius (r), following Laplace law P = 2.γ/r where γ is the surface tension. The pressure necessary to the re-expansion of a collapsed cell depends on its radius. Amato's team has showed in 2006 that within the same lung, several levels of alveolar aeration and thus several opening pressures coexist. The distribution of pressures was bimodal, with a peak around 30 cmH2O and a second around 40 cmH2O. Consequently, to allow complete re-expansion of atelectasis within a lung, it is necessary to apply a pressure at least equal to 30 cmH2O. The application of insufficient pressures cannot be expected to result in complete re-expansion of the lung, but rather in an increase in aeration of already aerated alveoli (whose radius is larger and whose opening pressure is much lower), what, in turn, can lead to over-distension. This is probably what can happen if the PEEP is increased without any previous ARM.

The application of an ARM can also lead to an overdistension phenomenon during a reduced period of time (20 to 30 seconds), contrary to the direct application of a high PEEP which could led to an overdistension lasting a much longer period of time (possibly several hours) and aggravated with each administration of a tidal volume (and thus several times per minute). Chronic lung exposure to overdistension phenomena can induce a disintegration of alveolar collagen fibers (volotrauma), leading to local inflammation (biotrauma) and systemic inflammation by releasing pro-inflammatory molecules (cytokines...) into the bloodstream and led to apoptosis in distant organs (kidney, digestive tract for example).

The optimization of mechanical ventilation requires the search for the optimal PEEP: insufficient, it cannot prevent atelectasis formation; too high, it would lead to alveolar overdistension. In current practice, the PEEP is determined arbitrary or following a stepwise titration, either by incremental or decremental steps. To date, scientific literature is not unequivocal concerning the use of ARMs and their safety. Thus, some teams prefer not to use ARMs and usually apply an upward PEEP level.

The concepts presented above are valid both in patients with healthy lungs and in patients with "sick" lungs, the archetype and most severe form of which is acute respiratory distress syndrome (ARDS), which is a frequent pathology in ICU (10 to 20% of patients admitted). Its definition is based on the Berlin criteria published in 2012. The morality varies between 30 and 40% depending on the severity of the respiratory impairment. Management of patients suffering from ARDS requires an optimization of oxygenation, which is based first of all on mechanical ventilation, whether invasive or not. Since the ARDS Network study published in 2000 in the New England Journal of Medicine, it has been globally accepted that tidal volumes should be reduced to no more than 6 mL/kg IBW. Ventilatory management is based on concepts of "baby lung" and "open lung". These concepts explain that it is mandatory to consider that the lung volume available for mechanical ventilation is very small compared to the healthy lung volume (baby lung) and that the reduction in tidal volume must be accompanied by adjustments to keep the lung "open", combating the formation of atelectasis by the use of sufficient PEEP and ARMs.

Far from this pulmonary pathology, any mechanically ventilated patient, whether in the ICU or operating theatre, must benefit from a protective strategy. Any inadequate adjustment of the ventilation parameters can lead to lung lesions induced by mechanical ventilation (VILI, Ventilator Induced Lung Injuries) and to lesions similar to those observed during ARDS.

We therefore propose to explore the impact on pulmonary aeration and ventilatory parameters of two different strategies of PEEP optimization during invasive mechanical ventilation in healthy lungs and ARDS ICU patients. This randomized controlled study would allow us to validate our hypotheses, depending on the respiratory mechanics and patient's pulmonary disease.The final aim of this study is to determine the effects of a strategy based on the application of an ARM followed by decremental PEEP titration, compared to an incremental PEEP strategy without ARM, on pulmonary and ventilatory physio-(patho)-logical parameters in ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* ICU patients with healthy lungs or lungs with Acute Respiratory Distress Syndrome (according to Berlin criteria) under mechanically invasive controlled ventilation (intubation or tracheotomy) in the early phase of admission (< 12h)
* Patient deeply sedated (BIS between 30 and 50) and possibly under neuromuscular blocking agents (TOF < 2/4 at the orbicular) in case of inspiratory efforts
* Patient hemodynamically stable with an optimized volemia using a monitoring system (see protocol).
* Consent to participate
* Patient benefiting from a Social Security Insurance

Exclusion Criteria:

* Refusal to participate to the proposed study
* Obese patient with BMI ≥ 35 kg.cm-2
* Significant hemodynamic instability defined as > 20% increase in catecholamine doses during the last hour, despite optimization of blood volume according to a pre-established protocol
* Contraindication to the use of the electro-impedance tomography technique

  * Thoracic lesions
  * Chest bandages
  * Pace-maker/Implantable defibrillator
* Contraindication to the performance of an alveolar recruitment maneuver

  * Major Emphysema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-09-12 (Actual); Primary Completion 2021-09-12 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Recruited lung volume at each PEEP level between the 2 strategies (incremental or decremental). | The last minute of each Peep Step
  : The main endpoint is the difference between the recruited lung volume measured by nitrogen washin-washout method at the end of each PEEP level (5th minute) with the basal value measured at the beginning of the protocol, between decremental and incremental stepwise PEEP titration

SECONDARY OUTCOMES:
Homogeneity of pulmonary aeration | The last minute of each Peep Step
  Evaluation by using the Electrical Impedance Tomography (EIT) - derived index Center of ventilation (CoV)
Homogeneity of pulmonary aeration | The last minute of each Peep Step
  Evaluation by using the Global Inhomogeneity index (GI) by electro-impedance tomography (EIT)
Regional impedance variation | Measurement during the last minute of each PEEP step
  Evaluation of regional impedance variation (TIV: Tidal Impedance Variation) by EIT
Atelectrauma | Measurement during the last minute of each PEEP step
  Assessement of atelectrauma (RVD: Regional Ventilation Delay) by EIT
Lung volume variations | Measurement during the last minute of each PEEP step
  Evaluation of lung volume variations by EIT (EELI : End Expiratory Lung Impedance)
Mechanical power delivered Mechanical power delivered | Measurement during the last minute of each PEEP step
  By using the formula : Power rs =RR⋅{ΔV² ⋅[1/2 ⋅ELrs +RR⋅((1+I:E) / (60⋅I:E) x Raw ]+ΔV⋅PEEP}. (Gattinoni, Intensive Care Medicine 2016)
Alveolar strain | Measurement during the last minute of each PEEP step
  Alveolar strain as assessed by TV/FRC where TV stands for tidal volume and FRC functional residual capacity.
Recruited lung volume | Measurement during the last minute of each PEEP step
  Evaluation of recruited lung volumes (Dellamonica, Intensive Care Medicine 2011)
Ventilatory dead space | Measurement during the last minute of each PEEP step
  Ventilatory dead space = Vd/Vt. Where Vd is the dead space volume and Vt is the tidal volume
Ventilatory parameters | Measurement during the last minute of each PEEP step
  Evaluation of the compliance = TV / (Pplat - PEEP) where TV stands for tidal volume, Pplat stands for Plateau Pressure and PEEP stands for Positive End-Expiratory Pressure
Ventilatory parameters | Measurement during the last minute of each PEEP step
  Evaluation of the driving pressure
Ventilatory parameters | Measurement during the last minute of each PEEP step
  Evaluation of the plateau pressure

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Godet, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU, Clermont-Ferrand, France